CLINICAL TRIAL: NCT04231721
Title: High Resolution Colonic Manometry in Relation to 3D-Transit Times in Healthy Controls.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Janne Ladefoged Fassov (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Janne Ladefoged Fassov, Principle investigator, MD, Ph.D., Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: 1-10-72-43-19; CIV-19-05-028726 (Other: Danish Competent Authority)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Colonic Motility
Keywords: Neurogastroenterology; Colonic motility; Manometry; High resolution colonic manometry; 3D-Transit system; Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy controls
  Interventions: Device: High Resolution Colonic Manometry and 3D-Transit system

INTERVENTIONS:
Device: High Resolution Colonic Manometry and 3D-Transit system — Measurement of colonic pressure changes and passage patterns in healthy.

SUMMARY:
Background: Within recent years, new methods for detailed assessment of gastrointestinal (GI) motility have been developed. Hence, the electromagnetic 3D-Transit system is a safe, non-invasive method for detailed description of GI motility. The system tracks the exact position of an ingested electromagnetic capsule through the entire GI tract and provides detailed information on both regional transit- and contraction patterns. High Resolution Colonic Manometry (HRCM) allows extremely detailed description of contraction patterns in the colon. The HRCM is however an invasive method, as the catheter is placed during colonoscopy. Before widespread use of capsule-based techniques (3D-Transit or others), the system needs to be validated by another method.

Study Objectives: The purpose of this study is to investigate weather pressure changes measured by HRCM correlate with passage patterns recorded by 3D-Transit. This has been assumed so far, but has never been further investigated.

Hypothesis: Movement of the electromagnetic 3D-Transit capsule within the colon correspond well with pressure changes determined with HRCM.

Materials and methods: HRCM and 3D-transit will be performed simultaneously in 20 healthy participants. A colonoscopy is performed to install the HRCM catheter and place two 3D-Transit capsules within the colon. For 24 hours, the participants lie in a bed in the research lab while pressure changes from the HRCM catheter are recorded and the 3D-Transit capsules are followed through the gastrointestinal system.

Perspectives: If data from the 3D-Transit technique correlate well with HRCM, the method provide a non-invasive alternative allowing detailed assessment of colonic motility.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Normal gastrointestinal function
* Psychologically able to give an informed content.

Exclusion Criteria:

* Known gastrointestinal disease
* Intake of medication with known effects on the movement patterns in the gastrointestinal system.
* Pregnancy and lactation
* Unable to follow the scheduled program in the trial due to mental illness or instability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All healthy individuals who meet the inclusion- and exclusion criteria can be enrolled in the study. The recruitment process will primarily take place through the Danish website "Forsoegspersoner.dk", which all Danish people have equal access to.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between pressure changes and passage patterns | 24 hours measurement
  Do the high amplitude propagating contraction patterns accessed with High Resolution Colonic Manometry occur simultaneously with the long fast antegrade movements determined with the 3D-Transit system.

SECONDARY OUTCOMES:
Distance of capsule movement and pressure changes | 24 hours measurement
  How do the length of a pressure change measured by High Resolution Colonic Manometry correlate with the distance covered in long fast antegrade movements determined with the 3D-Transit system (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Krogh, Professor, Study Director — Department of Hepatology and Gastroenterology, Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the possibility of data sharing.